CLINICAL TRIAL: NCT06470165
Title: Global Coronal Malalignment in Degenerative Lumbar Scoliosis and Priority-Matching Correction Technique to Prevent Postoperative Coronal Decompensation
Brief Title: Priority-Matching Correction Technique in Degenerative Lumbar Scoliosis
Acronym: PMCTDLS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: xuanwu_DLS
Record Dates: First submitted 2024-06-17; First posted 2024-06-24 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-01

CONDITIONS: Degenerative Lumbar Disease; Scoliosis; Degenerative Scoliosis
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DLS patients undergoing correction surgery in reference to our novel criteria (Experimental): Correcting deformity according to the priority-matching correction technique.
  Interventions: Procedure: Priority-matching correction technique in DLS
- DLS patients undergoing correction surgery in reference to Obeid classification (Other): Correcting deformity according to the standard proposed by Obeid and colleagues.
  Interventions: Procedure: Traditional correction technique in DLS

INTERVENTIONS:
Procedure: Priority-matching correction technique in DLS — For Type 1 global coronal malalignment (GCM), TL/L curve makes the primary contri- bution on C7PL shifting. First, inserting pedicle screws bilaterally. Second, aggressively decreasing the magnitude of TL/L curve. Third, moderately leveling L4 endplate to pull the fusion segments to the middle line with hand pressure on the convexity of TL/L curve. If the correctability of the key curve was limited, the correction of the minor curve would be con- vergent.
  For Type 2 GCM, LS curve makes the primary contribution on C7PL shifting. First, releasing LS curve from the concave side using facetectomy after screws inserted. Second, performing L4-5 or L5-S1 trans- foraminal lumbar interbody fusion (TLIF) from the con- vexity of the fractional curve, with cages inserted at the concave side to assist deformity correction. Third, compressing the convexity of LS to horizontalize L4 endplate, followed by moderate manipulative reduction of TL/L curve to adjust intraoperative coronal balance.
  Arms: DLS patients undergoing correction surgery in reference to our novel criteria
Procedure: Traditional correction technique in DLS — In concave coronal malalignment (CM), the correction of the main curve improves the CM, thus we can talk about convergent corrective objectives. The ability to correct the CM depends on the correctability of the main curve. The need of three-column osteotomies in order to obtain correction of CM depends on the location and flexibility of the main curve.
  The correction of convex CM depends on the correction of the lumbosacral curve. The correction strategy will depend on many factors including the driver of the deformity, which should always be fused, but also the degeneration and stiffness of the compensatory curve which can lead to more extended fusion. The need of three-column osteotomies depends mainly on the stiffness of the lumbosacral curve.
  Arms: DLS patients undergoing correction surgery in reference to Obeid classification

SUMMARY:
Surgical outcomes, including radiographic outcomes, patient-reported outcomes, postoperative complications, and revision surgery rates, were compared in patients with degenerative lumbar scoliosis (DLS) who underwent correction surgery with reference to our priority-matching correction technique and the standard reported by Obeid and colleagues. Our findings may provide tangible guidance for surgical decision-making in DLS.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of DLS based on radiography and previous medical record,
2. Age > 50 years

Exclusion Criteria:

1. Leg length discrepancy,
2. A history of spinal or pelvic surgery,
3. A history of neuromuscular diseases, arthritis or tumor.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-08-21 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Scoliosis Research Society-22 | One month, 3 months, 6 months, 1 year, and 2 years after surgery
  The 22-item SRS-22r questionnaire is specific to scoliosis-related patient-reported outcomes, and consists of 6 domains: function, pain, self-image, mental health, satisfaction, and subtotal, with each domain being scored from 1 to 5 where higher scores correspond to better patient outcomes.
Oswestry disability index | One month, 3 months, 6 months, 1 year, and 2 years after surgery
  The validated ODI is a self-administered questionnaire for evaluating back-specific functional disability, consisting of 10 items with scores from 0 to 5, and higher ODI indicates more severe disability.
Achievement of minimal clinically important difference | Two years after surgery
  A prespecified MCID of 10 points was used for the ODI. The minimum clinically important difference (MCID) values for the SRS-22r based on data from a Japanese cohort have previously been reported as follows: function = 0.90, pain = 0.85, self-image = 1.05, mental health = 0.70, and subtotal = 1.05.

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No